CLINICAL TRIAL: NCT01819441
Title: Azelnidipine vs Perindopril and Stratification of Blood Pressure Control Against Progress of Cerebral Small Vessel Diseases in Poststroke Patients (APPROVE):Multi-center Randomized Controlled Clinical Trial
Brief Title: Stratification of Blood Pressure Control Against Progress of Cerebral Small Vessel Diseases in Poststroke Patients
Acronym: APPROVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yining Huang (Other)
Responsible Party: Sponsor-Investigator, Yining Huang, chairman, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Peking University; APPROVE (Registry Identifier: Yining Huang)
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: cerebral small Vessel diseases, blood pressure,CCB, ACEI
MeSH Terms: conditions — Cerebral Small Vessel Diseases | interventions — azelnidipine; Perindopril; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Azelnidipine/Perindopril (Sham Comparator): Systole blood pressure controlled between 130 mmHg~140 mmHg(with or without hydrochlorothiazide).
  Interventions: Drug: Azelnidipine; Drug: Perindopril; Drug: hydrochlorothiazide
- Intensive Azelnidipine/Perindopril (Experimental): Systole blood pressure controlled below 130 mmHg(with or without hydrochlorothiazide).
  Interventions: Drug: Azelnidipine; Drug: Perindopril; Drug: hydrochlorothiazide

INTERVENTIONS:
Drug: Azelnidipine — 8mg or 16mg
  Other Names: BeiQi
Drug: Perindopril — 4mg or 8mg
  Other Names: YiTai
Drug: hydrochlorothiazide — 12.5mg or 25mg

SUMMARY:
A. the controlling of the blood pressure, especially the variation of blood pressure, can slow down the development of the small vessel disease.

B intensive BP control is more effective than normal control of blood pressure in slowing down the small vessel disease.

C drugs of Calcium Channel Blocker(CCB) and Angiotensin-Converting Enzyme Inhibitor(ACEI) have no significant difference in lowing the blood pressure and variability of blood pressure

DETAILED DESCRIPTION:
The selected patients were diagnosis of stroke caused by small vessel disease due to hypertension recently.

The patients had been divided into two groups by random principle and given ACEI or CCB separately for treatment. At the same time, given intensive or regular controlling of the blood pressure by stratified random. In the regular controlling group, the BP should be in the range of 130-139 mmHg and in the intensive controlling group, the BP should be below 130 mmHg. To the acute ischemic stroke patients who were accord with the lacunar infarction syndrome, it is rule to do the examination for exclusive selection of exclusion of hemodynamic dysfunction due to the artery stenosis ( stenosis >50%, the examination of intracranial artery was by the methods of Transcranial Doppler (TCD)/Magnetic Resonance Angiography(MRA)/Computed Tomographic Angiography(CTA)/Digital Subtraction Angiography(DSA), the examination of carotid artery was by the methods of colorful ultrasound / MRA/ CTA/ DSA ) at the baseline.

It should be proved of lacunar infarction by brain imaging. All patients had a MRI scan at the baseline and the beginning of the research, including T1-Weighted Imaging(T1W1),T2-Weighted Imaging(T2WI), T2-FLAIR, Diffusion-Weighted Imaging(DWI), Gradient-Recalled Echo(GRE) T2*, the Perfusion-Weighted Imaging(PWI) would complete conditionally (100 cases). The details should be followed by the instruction in the appendix.

Research about the variability of blood pressure: all patients show complete the examination of 24-hour blood-pressure monitor (at the baseline, the first month after the beginning, every three months and the end of the research), complete the head-up tilt test if conditionally ( at the baseline, each 3 months later and the end of the research ) The automatic regulation function of the small vessel should be evaluated if conditionally (the C02 reaction, TCD head-up tilt) and also the function of endothelium-derived relaxing of the brachial artery (at the baseline, each 3 months later and the end of the research) The reservation of the blood was for further research on genetic study.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral infarction within 10 days to 6 months.
* Clinical manifestation represented as lacunar infarction syndrome; without aphasia or disturbance of consciousness.
* Mini-Mental State Examination(MMSE)>24 and modified Rankin Score(mRS)≤3.
* History of hypertension, and need to be treated with drugs; patient who had been diagnosis hypertension or the first time with the diagnosis of this disease after the guideline of China 2010 (measurement of the BP in the seated posture of the up arm after having a rest for 5 minutes and was taken for three times and calculated the average result, make sure the difference of BP between right and left arm are not beyond the criteria of 20 mmHg and the right arm for consistence. The patients have different BP between both sides which the difference beyond 20 mmHg need to exam for the stenosis of subclavian artery.
* MRI confirm the lesion for lacunar infarction and be responsible for the clinical symptom located in the region of perforating artery and the diameter of the lesion is less than 20mm.
* The examinations of carotid artery and intracranial artery have excluded hemodynamic abnormalities due to artery stenosis ( stenosis >50%, the examination of intracranial artery was by the methods of TCD/ MRA/ CTA/ DSA, the examination of carotid artery was by the methods of colorful ultrasound / MRA/ CTA/ DSA ). The combination of thickness Intima media or plaque of the carotid artery without the hemodynamic dysfunction can be enrolled in this research.
* Informed consent was signed.

Exclusion Criteria:

* Hypertension diffcult to control, instantly over 220/ 120 mmHg.
* History of atrial fibrillation (Paroxysmal or sustained).
* History of heart infarction within 6 months.
* Stenosis above 50% or hemodynamic dysfunction in carotid and intracranial artery after examination.
* Unknown caused of brain infarction, like dissection vascular, Moyamoya disease, vasculitis, hereditary small angiopathy ( eg,Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leucoencephalopathy(CADASIL), FABRY, mitochondrial encephalopathy).
* Severe liver and renal disease. the definition of sever liver disease was Alanine aminotransferase(ALT) or Aspartate aminotransferase(AST) 4 times than the normal level, or the total bilirubin above 20 mmol/L, or cirrhosis. the definition of sever renal disease was stenosis of renal artery and dysfunction of renal (clearance rate of creatinine <60ml/min or serum creatinine >265mmol/L).
* History of hemorrhage.
* Active bleeding disease or clear coagulation disorders.
* Malignant neoplasm.
* Pregnancy.
* Severe organic diseases, expected lifetime was shorter than 2 years.
* Conditions contraindicated for CCB or ACEI, such as hyperpotassaemia (serum potassium >5.5mmol/L) or have the evidence proved allergic to both drugs.
* Eenrolled in another clinical trial in 30 days.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral Small Vessel Disease progressing | two years
  Area of WML increase more than 4% or Number of CMBs increase more than 2

CONTACTS AND LOCATIONS:
Overall Officials: Yining Huang, M.D., Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China